CLINICAL TRIAL: NCT06554847
Title: A Multi-Centered, Randomized, Double-Blinded, Placebo-Controlled Phase Ⅲ Clinical Trial to Evaluate the Efficacy and Safety of 611(Recombinant Humanized Anti-interleukin-4 Receptor Alpha IgG4 Monoclonal Antibody) When Used In Combination With Topical Corticosteroid Treatment (TCS) in Participants With Moderate to Severe Atopic Dermatitis.
Brief Title: Evaluation of 611 in Combination With Topical Corticosteroid in Participants With Moderate to Severe Atopic Dermatitis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSGJ-611-AD-III-02
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Dermatitis, Atopic; Eczema, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — entacapone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 611 interval 1+Topical Corticosteroid (Experimental): Participants will receive 611 according to established dosing interval 1. TCS will be initiated at Baseline in all patients and may be tapered or stopped, as needed, based on treatment response.
  Interventions: Drug: 611; Drug: Topical corticosteroid
- 611 interval 2+Topical Corticosteroid (Experimental): Participants will receive 611 according to established dosing interval 2. TCS will be initiated at Baseline in all patients and may be tapered or stopped, as needed, based on treatment response.
  Interventions: Drug: 611; Drug: Topical corticosteroid
- Placebo+Topical Corticosteroid (Placebo Comparator): Participants will receive Placebo according to according to established dosing intervals. TCS will be initiated at Baseline in all patients and may be tapered or stopped, as needed, based on treatment response.
  Interventions: Drug: Placebo; Drug: Topical corticosteroid

INTERVENTIONS:
Drug: 611 — subcutaneous injection
  Arms: 611 interval 1+Topical Corticosteroid; 611 interval 2+Topical Corticosteroid
Drug: Placebo — subcutaneous injection
  Arms: Placebo+Topical Corticosteroid
Drug: Topical corticosteroid — Topical

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group study to evaluate the safety and efficacy of 611 when used in combination with topical corticosteroid (TCS) treatment compared with placebo in combination with TCS treatment for moderate-to-severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults ages 18 to 75 years old when signing the informed consent.
* AD (according to Hanifin-Rajka Criteria) that had been present for at least 1 years before the screening visit.
* Moderate to Severe Atopic Dermatitis.
* Recent history of inadequate response to treatment with topical medications.

Exclusion Criteria:

* Participation in a prior 611 clinical study.
* Treatment with the following prior to the baseline visit: 1) Systemic corticosteroid or Immunosuppressants / Immunomodulators within 4 weeks or within 5 half-lives (if known), whichever is longer. 2) Monoclonal antibody within 5 half-lives (if known) or 4 months, whichever is longer. 3) Cell-depleting within 6 months.
* Treatment with a live (attenuated) vaccine within 2 months of the baseline visit or planned during the study.
* Serious or Uncontrolled diseases that may affect the safety of participants during the study period or hinder their completion of the study.
* Evidence of active acute or chronic hepatitis.
* History of malignancy within 5 years before the screening visit or currently.
* Pregnant or breastfeeding women, or women planning to become pregnant.
* Any history of vernal keratoconjunctivitis (VKC) and atopic keratoconjunctivitis (AKC).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-10-12 (Estimated); Study Completion 2026-08-16 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving EASI-75 (≥75% reduction from Baseline in EASI score) | Baseline to Week 16
Percentage of patients with an IGA score of 0 or 1 and a reduction ≥2-points from Baseline to Week 16. | Baseline to Week 16

SECONDARY OUTCOMES:
Percentage change in Pruritus Numerical Rating Scale (NRS) score from Baseline to Week 16 | Baseline to Week 16

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Shanghai Dermatology Hospital, Shanghai, Shanghai Municipality
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No